CLINICAL TRIAL: NCT02942758
Title: Randomized Phase II Trial With Safety run-in Phase Evaluating Low-dose AZA, ATRA and Pioglitazone Versus Standard Dose Azacitidine in Patients >=60 Years With AML Who Are Refractory to Standard Induction Chemotherapy
Brief Title: Low-dose AZA, Pioglitazone, ATRA Versus Standard-dose AZA in Patients >=60 Years With Refractory AML
Acronym: AML-ViVA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to financial reasons.
Sponsor: University Hospital Regensburg (Other)
Collaborators: Anticancer Fund, Belgium (Other); Celgene (Industry)
Responsible Party: Principal Investigator, Simone Thomas, Dr. med., University Hospital Regensburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMLSG26-16
Record Dates: First submitted 2016-10-18; First posted 2016-10-24 (Estimated); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; Pioglitazone; Tretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low-dose AZA / ATRA / Pioglitazone (Experimental): low-dose azacitidine (75 mg/d), ATRA, pioglitazone
  Interventions: Drug: low-dose Azacitidine; Drug: Pioglitazone; Drug: ATRA
- standard-dose AZA (Active Comparator): standard-dose azacitidine (75mg/m²/d)
  Interventions: Drug: standard-dose AZA

INTERVENTIONS:
Drug: low-dose Azacitidine — Azacitidine 75 mg/d s.c. for 7 days, repeated 28-day treatment cycle
  Other Names: Vidaza
  Arms: low-dose AZA / ATRA / Pioglitazone
Drug: Pioglitazone — Pioglitazone 45 mg p.o. continuously from day 1
  Other Names: Actos
  Arms: low-dose AZA / ATRA / Pioglitazone
Drug: ATRA — ATRA *45 mg/m² p.o. from day 1 to 28, 15 mg/m² from day 29 continuously; *this regimen will be chosen for the first dose to be evaluated.
  Other Names: All-trans-retinoic acid; Vesanoid
  Arms: low-dose AZA / ATRA / Pioglitazone
Drug: standard-dose AZA — Azacitidine 75 mg/m²/d s.c. for 7 days, repeated 28-day treatment cycle
  Other Names: Vidaza
  Arms: standard-dose AZA

SUMMARY:
Diagnosis: Acute myeloid leukemia refractory to intensive induction chemotherapy; Age ≥ 60 years, no upper age limit; Study drug: low-dose azacitidine, pioglitazone, ATRA; Safety Run-In Phase; randomized Phase II, open-label

* Safety Run-In Phase: Based on a 3 + 3 modified design, the tolerable dose of ATRA for the randomized phase II is defined.
* Phase II: Experimental Arm: low-dose azacitidine, pioglitazone, ATRA; Standard Arm: standard-dose azacitidine; in both arms patients can receive further cycles (with no limit to the number given) as long as clinically appropriate

ELIGIBILITY:
Inclusion Criteria:

1. Patients with confirmed diagnosis of acute myeloid leukemia (AML) who are refractory* to induction therapy and not eligible for further intensive induction therapy based on documented medical reasons (e.g. disease characteristics or patient characteristics), or
2. Patients with confirmed diagnosis of acute myeloid leukemia (AML) who are refractory* to induction therapy and not immediate candidates for allogeneic HSCT (bridge to transplant is allowed)

   *refractory to induction therapy is defined as no CR, no CRi and no PR (according to standard criteria, see Section 11.2.3) after at least one intensive induction therapy including at least 5 days of cytarabine 100-200 mg/m² continuously or an equivalent regimen with cytarabine with total dose not less than 500 mg/m² per cycle and at least 2 days of an anthracycline (e.g. daunorubicin, idarubicin).
3. Age ≥ 60; no upper age limit
4. ECOG performance status of ≤ 2 at screening
5. To control hyperleukocytosis or extramedullary involvement, medication with hydroxyurea is allowed up to 24h before start of study treatment. In case of hyperleukocytosis hydroxyurea should be given and start of study treatment should be delayed until leukocyte counts are < 20 x 10^9/L.
6. Female subjects of childbearing potential* may participate, providing they meet the following conditions:

   * Have a negative pregnancy test (serum or urine with a sensitivity of at least 25 mIU/mL; local laboratory) within 72 hours prior to starting study therapy. They must agree to ongoing pregnancy testing during the course of the study, and after end of study therapy. This applies even if the subject practices true abstinence** from heterosexual contact.
   * Agree to practice true abstinence** from heterosexual contact (which must be reviewed on a monthly basis) or agree to use, and be able to comply with two effective methods of contraception (e.g., oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) without interruption during the study therapy (including dose interruptions), and for 3 months after discontinuation of study drugs.

     * A female subject of childbearing potential (FCBP) is a female who: 1) has achieved menarche at some point 2) has not undergone a hysterectomy or bilateral oophorectomy or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (ie, has had menses at any time in the preceding 24 consecutive months).

       * True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (eg, calendar, ovulation, symptothermal, postovulation methods) and withdrawal are not acceptable methods of contraception.
7. Male patients with a female partner of childbearing potential must agree to abstain from sexual intercourse or to the use of at least two effective contraceptive methods (e.g., synthetic condoms with spermicide, etc) at screening and throughout the course of the study and should avoid fathering a child during the course of the study and for 3 months following the last study treatment.
8. Signed written informed consent.

Exclusion Criteria:

1. Known or suspected hypersensitivity to the study drugs and/or any excipients
2. Patients with acute promyelocytic leukemia exhibiting t(15;17)(q22;q12); PML-RARA, or with variant translocations
3. Acute myeloid leukemia (AML) with isocitratdehydrogenase (IDH) 1 or 2 mutations if results are available from the central AMLSG reference laboratories
4. ECOG performance status > 2
5. Inadequate cardiac, hepatic and/or renal function at Screening Visit defined as:

   1. heart failure NYHA II-IV
   2. unstable angina pectoris
   3. total bilirubin, ALT, AST > 2.5 x upper normal serum level
   4. Creatinine > 1.5 x upper normal serum level
6. Active central nervous system involvement
7. Uncontrolled infection
8. Uncontrolled diabetes mellitus
9. Patients with a "currently active" second malignancy requiring active therapy other than non-melanoma skin cancers (except for hormonal/antihormonal treatment, e.g. in prostate or breast cancer)
10. Patients with "currently active" bladder cancer or bladder cancer in their history, patients with risk factors for bladder cancer (e.g. exposure to aromatic amines or heavy tobacco smoker), or macrohematuria of unknown origin
11. Severe neurological or psychiatric disorder interfering with ability of giving an informed consent
12. Known or suspected active alcohol or drug abuse
13. Known positive for HIV, active HBV or HCV infection
14. No consent for registration, storage and processing of the individual disease characteristics and course as well as information of the family physician and/or other physicians involved in the treatment of the patient about study participation.
15. Treatment with any other clinical study drug within 14 days before the first administration of the investigational drugs or at any time during the study
16. Breast feeding woman or women with a positive pregnancy test at Screening Visit
17. Male patients with a female partner of childbearing potential not willing to abstain from sexual intercourse or to the use of at least two effective contraceptive methods (e.g., synthetic condoms with spermicide, etc) at screening and throughout the course of the study and for 3 months following the last study treatment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
overall Survival | 3 years

SECONDARY OUTCOMES:
complete remission (CR) rate | 3 years
complete remission with incomplete blood count recovery (CRi) rate | 3 years
partial remission (PR) rate | 3 years
hematological improvement (HI) rate | 3 years
cumulative incidence of relapse (CIR) | 3 years
cumulative incidence of death (CID) | 3 years
cumulative incidence of relapse event free survival (EFS) | 3 years
event free survival (EFS) | 3 years
Quality of Life (QLQ-C30) | 3 years
Incidence and intensity of adverse events (AEs) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Simone Thomas, Dr., Principal Investigator — University Hospital Regensburg
Locations (1):
- University Hospital Regensburg, Regensburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Klobuch S, Steinberg T, Bruni E, Mirbeth C, Heilmeier B, Ghibelli L, Herr W, Reichle A, Thomas S. Biomodulatory Treatment With Azacitidine, All-trans Retinoic Acid and Pioglitazone Induces Differentiation of Primary AML Blasts Into Neutrophil Like Cells Capable of ROS Production and Phagocytosis. Front Pharmacol. 2018 Nov 27;9:1380. doi: 10.3389/fphar.2018.01380. eCollection 2018. PMID 30542286